CLINICAL TRIAL: NCT06483230
Title: A Pilot Study on Tolerance and Ease of Implementation of Intensive Visual Stimulation (IVS3) in Daily Practice for Upper Limb Motor Recovery in Outpatient Rehab Center
Brief Title: Implementation of IVS3 for Upper Limb Motor Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Dessintey Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-04027379
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Neglect, Hemispatial; Stroke, Cardiovascular; Mirror Movement; Motor Activity
MeSH Terms: conditions — Perceptual Disorders; Myocardial Infarction; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hemi-spatial Neglect (Experimental): Individuals with stroke with hemi-spatial neglect as identified on the star cancellation and line bisection tests.
  Interventions: Device: Intensive Visual Stimulation Device
- No hemi-spatial neglect (Active Comparator): Individuals with stroke without hemi-spatial neglect as identified on the star cancellation and line bisection tests.
  Interventions: Device: Intensive Visual Stimulation Device

INTERVENTIONS:
Device: Intensive Visual Stimulation Device — The therapist installs the patient in front of the device. First, patient puts the healthy side on the table and the therapist records several movements. The software of the device flips the video in order to create a mirrored image of the movement (pretty close to the mirror therapy approach). When all the movements are recorded, patient installs the affected side on the table and the screen is placed over the hand. Likewise, patient has the impression the hand is moving again. Thanks to this action observation principle, therapist can encourage the patient in trying to move again and increase brain plasticity.
  Other Names: IVS3 (model number 2022.02.IVS3.013)

SUMMARY:
This study measures participant satisfaction and upper extremity function in outpatients with chronic stroke when exposed to the IVS3 device. Investigators hypothesize that treatment with the IVS3 device will be feasible and tolerable for use in the outpatient setting.

DETAILED DESCRIPTION:
This study will investigate the implementation of the intensive visual stimulation three (IVS3) device in the outpatient rehabilitation setting. This is a phase I/II open label study that will assess participant satisfaction and upper extremity function in outpatients with chronic stroke (10 with hemi spatial neglect and 15 without), when exposed to IVS3 for 30 minutes and conventional treatment for 15 minutes, across 12 sessions in 4-6 weeks at Weill Cornell medicine outpatient rehabilitation (single site).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. English speaking
3. History of ischemic or hemorrhagic stroke ≥ 6 months prior to study enrolment
4. FMA-UE: 20 < x < 50 (moderate impairments)
5. With or without hemi spatial neglect

Exclusion Criteria:

1. Spasticity or increased tone with MAS ≥3 in the upper extremity
2. Unable to communicate effectively or provide informed consent
3. Significant visual impairments
4. Concurrent occupational therapy being received outside of the study
5. Pregnant or incarcerated individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Mean number of sessions attended | 12 treatment sessions over 4-6 weeks.
  The primary outcome measure is defined as the mean number of sessions attended of the planned twelve visits. Min 0, Max 12.
Number of serious adverse events | 12 treatment sessions over 4-6 weeks.
  The primary outcome for safety is defined as the number of serious adverse events that occur while using the IVS3 device.

SECONDARY OUTCOMES:
Mean Client Satisfaction Questionnaire-8 | Post- treatment (Weeks 6-11, Visit 14), 3 months post-treatment (Weeks 18-23, Visit 15)
  Feasibility. This tool is a self-report measure participant satisfaction with the intervention. Scored 8-32 with higher scores indicating greater satisfaction.
Mean System Usability Scale (SUS) | Post- treatment (Weeks 6-11, Visit 14), 3 months post-treatment (Weeks 18-23, Visit 15)
  Feasibility. This tool is a subjective therapist usability measure assessing satisfaction with implementation of the intervention. It is a 10 item likert scale, scored 0-100, with higher scores indicating greater satisfaction.

OTHER OUTCOMES:
Mean Star Ratio on Star Cancellation Test | Baseline (Week 1, Visit 1), Post- treatment (Weeks 6-11, Visit 14), 3 months post-treatment (Weeks 18-23, Visit 15)
  Screening tool to detect unilateral spatial neglect. The maximum score that can be achieved on the test is 54 points (56 small stars in total minus the 2 used for demonstration). A cutoff of < 44 indicates the presence of USN. A Laterality Index or Star Ratio can be calculated from the ratio of stars cancelled on the left of the page to the total number of stars cancelled. Scores between 0 and 0.46 indicate USN in the left hemispace. Scores between 0.54 and 1 indicate USN in the right hemispace
Mean Distance from Midpoint on Line Bisection | Baseline, Post- treatment, 3 months post-treatment.Baseline (Week 1, Visit 1), Post- treatment (Weeks 6-11, Visit 14), 3 months post-treatment (Weeks 18-23, Visit 15)
  Screening tool to detect unilateral spatial neglect. Patients are asked to place a mark with a pencil (with their preferred or unaffected hand) through the center of a series of 18 horizontal lines on an 11x 8.5-inch page. The test is scored by measuring the deviation of the bisection from the true center of the line. A deviation of more than 6 mm from the midpoint indicates USN. Omission of two or more lines on one half of the page indicates USN.
Mean Change from baseline Fugl-Meyer Upper Extremity Assessment (FMAUE) | Baseline (Week 1, Visit 1), Post- treatment (Weeks 6-11, Visit 14), 3 months post-treatment (Weeks 18-23, Visit 15)
  Assessment of upper extremity motor function. Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform; 1=performs partially; and 2=performs fully. Score ranges from 0-66 for the upper extremity (22 items).
Mean Change from baseline Action Research Arm Test (ARAT) | Baseline (Week 1, Visit 1), Post- treatment (Weeks 6-11, Visit 14), 3 months post-treatment (Weeks 18-23, Visit 15)
  The Action Research Arm Test (ARAT) is an evaluative measure to assess specific changes in limb function among individuals who sustained cortical damage resulting in hemiplegia. The ARAT consists of 19 items grouped into four subscales: grasp, grip, pinch, and gross movement.The ARAT is scored on a four-level ordinal scale (0-3). 0 = can not perform any part of the test,
  1 = performs the test partially, 2 = completes the test, but takes abnormally long time, 3 = performs the test normally. Total score ranges from 0 to 57, with the lowest score indicating that no movements can be performed, and the upper score indicating normal performance.
Mean change from baseline numeric pain rating scale (NPRS) | Baseline (Week 1, Visit 1), Post- treatment (Weeks 6-11, Visit 14), 3 months post-treatment (Weeks 18-23, Visit 15)
  The NPRS measures the subjective intensity of pain. The NPRS is an 11-point scale scored from 0-10:
  1) "0" = no pain, 2) "10" = the most intense pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Stilling, MD,MS, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, 525 E. 68th St, Baker Pavilion, F-2106, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after de-identification (text, tables, figures).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 24 months following study publication
Access Criteria: Investigators whose proposed use of data has been approved by an independent review committee for individual participant data meta-analyses. Data will be available 2 years following study publication.